CLINICAL TRIAL: NCT03841383
Title: Study to Investigate the Association Between Coronary Flow Reserve and BH4 Levels in Patients With High Cardiovascular Risk
Brief Title: Association Between Coronary Flow Reserve and BH4 Levels in High CV Risk
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Servier (Industry)
Responsible Party: Principal Investigator, Prof. Paolo G Camici MD FACC, Professor of Cardiology, IRCCS San Raffaele
Other Study IDs: CFRBH4_IT1
Record Dates: First submitted 2019-01-25; First posted 2019-02-15 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Hypertension,Essential
MeSH Terms: conditions — Essential Hypertension | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy controls
  Interventions: Diagnostic Test: Echo stress dipyridamole
- Hypertensive patients
  Interventions: Diagnostic Test: Echo stress dipyridamole

INTERVENTIONS:
Diagnostic Test: Echo stress dipyridamole — Echo stress dipyridamole
  Other Names: Blood sample

SUMMARY:
To determine if there is a relationship between coronary flow reserve (CFR) and platelet/plasma BH2 and BH4 levels in patients with high cardiovascular risk .

DETAILED DESCRIPTION:
Primary parameter :

relationship between coronary flow reserve (CFR) and platelet/plasma BH2 and BH4 levels in patients with hypertension and concomitant cardiovascular risk factors.

Secondary parameter:

Levels of cGMP in platelets.

4. Study design

Three parallel groups of patients (n=15 per group):

* Group 1 with normal coronary flow reserve (CFR ≥2.5)
* Group 2 with reduced coronary flow reserve (CFR≤2.0)

  o Group 3 control subjects (without a high risk profile according to ESC score chart http://www.heartscore.org. ) matched for age (between 40 and 80 years of age)
* and gender. 1/3 enrolled patients must be diabetic (Type2 diabetes)

ELIGIBILITY:
Inclusion Criteria:

* o men and women (females of childbearing potential must be using highly effective contraceptive precautions such as implants, injectables, combined oral contraceptives, intrauterine devices, sexual abstinence or vasectomised partner)

  * Females of childbearing potential or within two years from the menopause must have a negative urine pregnancy test
  * between 40 and 80 years of age
  * documented history of hypertension
  * smokers/non smokers R
  * type 2 diabetes R
  * Moderate to severe kidney disease (GFR >30 and <60 ml/min/1.73m2 (estimated MDRD) R
  * Hypercholesterolemia R
  * Receiving an optimal standard antihypertensive treatment for at least 6 months, stable for at least 15 days
  * All other concomitant treatments stabilized at least for the preceding 15 days
  * Able to give written informed consent

Exclusion Criteria:

* o Females of childbearing potential not using highly effective contraceptive precautions

  * Patients with obstructive (>50% diameter reduction) CAD on the LAD (based on invasive angiography or coronary CTA) or with evidence of previous myocardial infarction or history of revascularization in the LAD territory.
  * CAD on the RCA or CX with diameter reduction > 50% (based on invasive angiography or coronary CTA) , either native or revascularized (stent)
  * Patients with infectious disease and/or chronic inflammatory diseases
  * Epicardial coronary arteries spasm
  * Patients with severe valve disease and/or significant left ventricular wall motion abnormalities
  * Patients under treatment with non-selective beta blockers including propranolol, nadolol, pindolol, labetalol, penbutolol, sotalol, carvedilol, and timolol.
  * Contraindications to dipyridamole infusion: asthma, bronchospasm, previous < 24 hours ingestion of phylline derivatives (tea, coffee, cola, xanthines and chocolate) sick sinus syndrome, advanced AV block (second and third degree), systolic blood pressure < 90 mmHg, cerebral ischemia, severe sinus bradycardia (heart rate <40/min), use of dipyridamole during the last 24 h, severe atherosclerotic lesions of extracranial artery >75%.
  * Acute treatment or treatment for acute diseases
  * Patients receiving steroidal anti-inflammatory drugs, dietary supplements of folic acid, or antioxidant vitamins.
  * Any condition that may prevent the pt to give informed consent , enter the study or bias the results.
  * Participating into other studies

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Symptomatic (angina symptoms both typical and atypical ) patients referred to the hospital with hypertension plus risk factors: diabetes, hypercholesterolemia, smoking, chronic renal failure
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-07-10 (Actual)

PRIMARY OUTCOMES:
BH2 and BH4 levels (ng/ml) in plasma and platelets | 1 week
  Blood samples will be withdrawn and subsequently analyzed to assess biopterins BH4 and BH2 ng/mL concentration in plasma and platelets Each will be determined separately from the same sample, by high-performance liquid chromatography followed by serial electrochemical and fluorescent detection.
Coronary Flow Reserve (CFR) Trans Thoracic Doppler Echocardiography | 1 week
  Measurement of coronary flow reserve of the left anterior descending coronary artery will be carried out with transthoracic Doppler Echocardiography (TDE) and dipyridamole stress. CFR will be calculated as the ratio between stress and resting flow velocity (cm/sec)
Relationship between coronary flow reserve (CFR) and platelet/plasma BH2 and BH4 levels. | 1 week
  Simple regression analysis or logistic regression will be used to test the relationship between CFR and biopterins values in plasma and platelets.

SECONDARY OUTCOMES:
Levels of cGMP in platelets | 1 week
  Comparison of levels of cGMP in platelets among normals, patients with normal CFR and patients with reduced CFR

CONTACTS AND LOCATIONS:
Overall Officials: Paolo G Camici, MD, Principal Investigator — IRCCS Ospedale San Raffaele
Locations (2):
- Italy (2):
  - ASST Papa Giovanni XXIII, Bergamo
  - IRCCS Ospedale San Raffaele, Milan

IPD SHARING:
Plan to Share IPD: Undecided